CLINICAL TRIAL: NCT02401880
Title: Effects of Linagliptin in Addition to Empagliflozin on Islet Cell Physiology and Metabolic Control in Patients With Type 2 Diabetes Mellitus on Stable Metformin Treatment
Brief Title: Effects of Linagliptin in Addition to Empagliflozin on Islet Cell Physiology
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Profil Institut für Stoffwechselforschung GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: EMLIN-001
Record Dates: First submitted 2014-12-11; First posted 2015-03-30 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2016-02

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Linagliptin; empagliflozin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Empagliflozin plus Linagliptin (Active Comparator): Linagliptin 5mg to be adminstered for 30 days in T2DM patients on stable metformin and Empagliflozin
  Interventions: Drug: Linagliptin; Drug: Empagliflozin
- Empagliflozin plus Placebo (Placebo Comparator): Placebo to be adminstered for 30 days in T2DM patients on stable metformin and Empagliflozin
  Interventions: Other: Placebo; Drug: Empagliflozin
- Empagliflozin (Other): Empagliflozin 25mg will be adminstered for 30 days in T2DM patients
  Interventions: Drug: Empagliflozin

INTERVENTIONS:
Drug: Linagliptin — 22 subjects will receive Linagliptin for 30 days
  Other Names: Trajenta
  Arms: Empagliflozin plus Linagliptin
Other: Placebo — 22 subjects will receive Placebo for 30 days
  Arms: Empagliflozin plus Placebo
Drug: Empagliflozin — 44 subjects will receive Empagliflozin for 60 days
  Other Names: Jardiance

SUMMARY:
The primary aim of this exploratory mechanistic study is to investigate the effects of Empagliflozin and Linagliptin on alpha- and beta cell physiology in T2DM patients.

This study aims to evaluate the effect of the DPP-IV inhibitor linagliptin (as compared to placebo) in addition to the SGLT-2 inhibitor empagliflozin on pancreatic alpha and beta cell function, as well as several markers of metabolic control.

DETAILED DESCRIPTION:
This study will be performed as a multi-center study which includes 2 centres. 44 subjects with T2DM are to be included according to the defined in- and exclusion criteria.

Subjects has to be on a stable metformin therapy and will receive in a first step empagliflozin for 30 days. Both therapies (metformin and empagliflozin) will be continued for another 30 days and subjects will be randomized to receive in addition Linagliptin or Placebo for 30 days.

Subjects will come for two inhouse periods to their corresponding study center and will undergo an hyperglycaemic clamp test as well as a Meal test in each of the periods.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subject with diabetes mellitus type 2
2. Diabetes mellitus type 2 on stable treatment with metformin (daily dose at least 1000 mg) for at least 6 months
3. HbA1c 7.0%-9.9%, both inclusive
4. Diabetes duration of at least 24 months)

Exclusion Criteria:

1. History of diabetes mellitus type 1
2. GFR (as calculated by the Cockcroft-Gault equation) < 60 ml/min at Screening
3. Systolic blood pressure outside the range of 100-160 mmHg or diastolic blood pressure above 95 mmHg at Screening

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2015-05; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
• Change in glucagon release (AUC0-180 min) during Liquid Meal Test (LMT) from V3 to V4 between the two treatment groups (Linagliptin vs. placebo) | 30 days

SECONDARY OUTCOMES:
• Change in glucagon release (AUC0-180 min) during LMT from V2 to V3 during treatment with Empagliflozin (V2 vs. V3) | 30 days

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - Profil Mainz GmbH & Co. KG, Mainz
  - Profil Institut für Stoffwechselforschung GmbH, Neuss